CLINICAL TRIAL: NCT06951490
Title: Assessing Negative PillSense™ for Safe Discharge in Patients With Positive Hemoccult and/or Unexplained Anemia
Brief Title: PillSense Use in Anemia and Hemoccult
Acronym: PillSense™
Status: Enrolling by invitation | Type: Observational
Sponsor: AdventHealth (Other)
Collaborators: EnteraSense Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 2232176
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-04

CONDITIONS: Occult Gastrointestinal Bleeding; Upper Gastrointestinal Bleeding (UGIB)
Keywords: PillSense; Upper Gastrointestinal Bleeding; GI Bleed Detection; Positive Hemoccult; Capsule Endoscopy; Non-invasive Diagnostics; Real-time GI Bleed Detection
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Hospitalized Patients Undergoing PillSense™ Testing: This group includes hospitalized adult patients who have been referred to gastroenterology services for unexplained anemia and/or a positive fecal occult blood test (hemoccult) in the absence of overt gastrointestinal bleeding (e.g., no melena, hematemesis, or hematochezia). All participants will ingest the PillSense™ capsule.
  Interventions: Device: PillSense™

INTERVENTIONS:
Device: PillSense™ — The PillSense™ System is a prescription only device consisting of a reusable receiver and single-use ingestible capsule, intended to be used for the detection of blood in the upper gastrointestinal tract.

SUMMARY:
In this study, participants will be offered a PillSense™ capsule, a small capsule to swallow, which can detect the presence of blood in the upper digestive tract within about 10 minutes. The results of this capsule test will not alter the current care plan but will help us assess whether PillSense™ can be used in the future as a standalone test to determine if it is safe for patients to be discharged with anemia or a positive stool test without other signs of gastrointestinal bleeding. This study aims to collect data that will help determine if the PillSense™ capsule could one day reduce the need for more invasive procedures while hospitalized, like endoscopy, and ensure safe patient discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to provide informed consent
* Hospitalized patients who have been referred to the gastroenterology service for:

A positive hemoccult (fecal occult blood test) and/or Anemia, In the absence of overt gastrointestinal bleeding - Overt gastrointestinal bleeding is defined as the presence of: Melena (black, tarry stools) Hematochezia (bright red blood per rectum) Hematemesis (vomiting blood)

Exclusion Criteria:

* Hemodynamic instability, defined as:

Systolic blood pressure < 90 mm Hg Pulse > 120 bpm

* Presence of overt gastrointestinal bleeding (melena, hematochezia, or hematemesis)
* Conditions that might contraindicate use of an ingestible capsule, such as:

Dysphagia or odynophagia Swallowing disorder Altered mental status Zenker's diverticulum Crohn's disease Previous GI surgery Suspected ileus or bowel obstruction GI perforation GI motility disorders (e.g., esophageal dysmotility, gastroparesis)

- Known upper GI pathology, such as: Esophageal or gastric cancer Recent upper GI ulcer bleeding (within 3 months) Recent upper GI procedures or surgeries

* Presence of a cardiac implantable electronic device (CIED)
* Pregnant or lactating women
* Planned MRI before capsule excretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of hospitalized adult patients who have been referred to the gastroenterology service for evaluation of unexplained anemia and/or a positive fecal occult blood test (hemoccult) in the absence of overt gastrointestinal bleeding. These patients represent a group commonly subjected to diagnostic endoscopy despite the often-low diagnostic yield of such procedures.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Negative PillSense™ Result in Predicting Safe Discharge | 24 hours
  To measure the percentage of participants with a negative Pillsense™ result who are safely discharged from the hospital without requiring urgent endoscopic intervention or experiencing adverse events during their hospitalization.

SECONDARY OUTCOMES:
False Negative Rate of PillSense™ | During hospitalization (up to 72 hours after capsule ingestion)
  Rate at which a negative PillSense™ results fail to detect clinically significant upper gastrointestinal bleeding later confirmed by endoscopy.
Timing of Endoscopic Intervention | 24-72 hours
  The average number of hours between taking the PillSense capsule and having an upper endoscopy, compared between patients with positive and negative PillSense results, to see if test results affect how quickly endoscopy is done.
Length of Hospital Stay | 24-72 hours
  Measure the average hospital length of stay (in days) between patients with positive and negative PillSense™ results to evaluate whether test outcome is associated with differences in duration of hospitalization.
30-Day Readmission Rate | 30 days post-discharge
  Rate of readmission within 30 days post-discharge between patients with positive and negative PillSense™ results.
30-Day Mortality | 30 days post-discharge
  All-cause mortality rate between patients with positive and negative PillSense™ results.

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing information from this study.

REFERENCES:
- [Background] Yung DE, Plevris JN, Koulaouzidis A. Short article: Aspiration of capsule endoscopes: a comprehensive review of the existing literature. Eur J Gastroenterol Hepatol. 2017 Apr;29(4):428-434. doi: 10.1097/MEG.0000000000000821. PMID 28253209
- [Background] Nemeth A, Wurm Johansson G, Nielsen J, Thorlacius H, Toth E. Capsule retention related to small bowel capsule endoscopy: a large European single-center 10-year clinical experience. United European Gastroenterol J. 2017 Aug;5(5):677-686. doi: 10.1177/2050640616675219. Epub 2016 Oct 16. PMID 28815031
- [Background] Rondonotti E, Soncini M, Girelli C, Ballardini G, Bianchi G, Brunati S, Centenara L, Cesari P, Cortelezzi C, Curioni S, Gozzini C, Gullotta R, Lazzaroni M, Maino M, Mandelli G, Mantovani N, Morandi E, Pansoni C, Piubello W, Putignano R, Schalling R, Tatarella M, Villa F, Vitagliano P, Russo A, Conte D, Masci E, de Franchis R; AIGO, SIED and SIGE Lombardia. Small bowel capsule endoscopy in clinical practice: a multicenter 7-year survey. Eur J Gastroenterol Hepatol. 2010 Nov;22(11):1380-6. doi: 10.1097/MEG.0b013e3283352ced. PMID 20173646
- [Background] Lim YJ, Lee OY, Jeen YT, Lim CY, Cheung DY, Cheon JH, Ye BD, Song HJ, Kim JS, Do JH, Lee KJ, Shim KN, Chang DK, Park CH, Jang BI, Moon JS, Chun HJ, Choi MG, Kim JO; Korean Gut Image Study Group. Indications for Detection, Completion, and Retention Rates of Small Bowel Capsule Endoscopy Based on the 10-Year Data from the Korean Capsule Endoscopy Registry. Clin Endosc. 2015 Sep;48(5):399-404. doi: 10.5946/ce.2015.48.5.399. Epub 2015 Sep 30. PMID 26473123
- [Background] Liao Z, Gao R, Xu C, Li ZS. Indications and detection, completion, and retention rates of small-bowel capsule endoscopy: a systematic review. Gastrointest Endosc. 2010 Feb;71(2):280-6. doi: 10.1016/j.gie.2009.09.031. PMID 20152309
- [Background] Fernandez-Urien I, Carretero C, Gonzalez B, Pons V, Caunedo A, Valle J, Redondo-Cerezo E, Lopez-Higueras A, Valdes M, Menchen P, Fernandez P, Munoz-Navas M, Jimenez J, Herrerias JM. Incidence, clinical outcomes, and therapeutic approaches of capsule endoscopy-related adverse events in a large study population. Rev Esp Enferm Dig. 2015 Dec;107(12):745-52. doi: 10.17235/reed.2015.3820/2015. PMID 26671587
- [Background] Rezapour M, Amadi C, Gerson LB. Retention associated with video capsule endoscopy: systematic review and meta-analysis. Gastrointest Endosc. 2017 Jun;85(6):1157-1168.e2. doi: 10.1016/j.gie.2016.12.024. Epub 2017 Jan 6. PMID 28069475
- [Background] Sachdev MS, Leighton JA, Fleischer DE, Heigh RI, Hara AK, Post JA, Erickson PJ, Sharma VK. A prospective study of the utility of abdominal radiographs after capsule endoscopy for the diagnosis of capsule retention. Gastrointest Endosc. 2007 Nov;66(5):894-900. doi: 10.1016/j.gie.2007.06.066. PMID 17963875
- [Background] Akiki K, Mahmoud T, Alqaisieh MH, Sayegh LN, Lescalleet KE, Abu Dayyeh BK, Wong Kee Song LM, Larson MV, Bruining DH, Coelho-Prabhu N, Buttar NS, Sedlack RE, Chandrasekhara V, Leggett CL, Law RJ, Rajan E, Gleeson FC, Alexander JA, Storm AC. A novel blood-sensing capsule for rapid detection of upper GI bleeding: a prospective clinical trial. Gastrointest Endosc. 2024 May;99(5):712-720. doi: 10.1016/j.gie.2023.11.051. Epub 2023 Dec 6. PMID 38065512
- [Background] Niv E, Elis A, Zissin R, Naftali T, Novis B, Lishner M. Iron deficiency anemia in patients without gastrointestinal symptoms--a prospective study. Fam Pract. 2005 Feb;22(1):58-61. doi: 10.1093/fampra/cmh705. Epub 2005 Jan 11. PMID 15644385
- [Background] Stray N, Weberg R. A prospective study of same day bi-directional endoscopy in the evaluation of patients with occult gastrointestinal bleeding. Scand J Gastroenterol. 2006 Jul;41(7):844-50. doi: 10.1080/00365520500495789. PMID 16785199
- [Background] Urquhart J, Eisen G, Faigel DO, Mattek N, Holub J, Lieberman DA. A closer look at same-day bidirectional endoscopy. Gastrointest Endosc. 2009 Feb;69(2):271-7. doi: 10.1016/j.gie.2008.04.063. Epub 2008 Aug 23. PMID 18725159
- [Background] Lin K, Linn S, Ramai D, et al. Clinical Features and Outcomes in Hospitalized Patients With Positive FOBT Undergoing Bidirectional Endoscopy - A Single-Center Experience: 2736. American Journal of Gastroenterology. 2018;113(Supplement):S1523. doi:10.14309/00000434-201810001-02735
- [Background] Barakat M, Aloreidi K, Gujjula S, et al. Overutilization of Fecal Occult Blood Test in the Acute Hospital Setting and its Impact on Clinical Management and Outcomes. Gastroenterology. 2020;159(2):e21-e22. doi:10.1053/j.gastro.2020.06.059